CLINICAL TRIAL: NCT04281641
Title: Gene Expression Assays and 68 Ga-Affibody HER-2 Imaging PET in Predicting Response to Treatment With Trastuzumab and Pertuzumab Before Surgery in Chinese Patients With HER2 Positive Breast Cancer
Brief Title: Markers to Evaluate the Efficacy of PH-based Regimen as a Neoadjuvant Therapy for Operable HER2 Positive Breast Cancer
Acronym: PHC-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Department of Breast Surgery Vice President, Cancer Hospital, Fudan University, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCHBCC-NO28
Record Dates: First submitted 2020-02-12; First posted 2020-02-24 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCHP (Experimental): Neoadjuvant Therapy (Cycles 1-7):
  Cycle 1: Pertuzumab (840mg loading dose, 420mg maintenance dose) + Trastuzumab (8mg/kg loading dose, 6-mg/kg maintenance dose) Cycle 2-7: Pertuzumab (840mg loading dose, 420mg maintenance dose) + Trastuzumab (8mg/kg loading dose, 6-mg/kg maintenance dose) + followed by carboplatin at target area under the plasma concentration-time curve (AUC) 6 and docetaxel at a starting dose of 75 mg/m2 then to 60mg/m2 (q3w).
  Adjuvant Therapy:patients would complete 1 year of PH-based regimen in the adjuvant setting.
  Patients are assessed by [18F]Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) and 68Ga-Affibody HER-2 Imaging PET. Besides, the changes of biomarkers would be examined by gene sequencing and organoid drug sensitivity test.
  Interventions: Diagnostic Test: TCHP

INTERVENTIONS:
Diagnostic Test: TCHP — Drug: Trastuzumab 8 mg/kg loading dose, then 6 mg/kg every 3 weeks, IV Other Name: Herceptin
  Drug: Pertuzumab 840 mg as a loading dose, then 420 mg every 3 weeks, IV Other Name: Perjeta
  Drug: carboplatin at target area under the plasma concentration-time curve (AUC) 6
  Drug: docetaxel at a starting dose of 75 mg/m2 then to 60mg/m2 (q3w).
  All study drugs were administered intravenously.
  Procedure: 18-FDG-PET and 68 Ga-Affibody HER-2 Imaging PET will be performed at baseline, on day 15 and before surgery
  Genomic alterations (mutations/somatic rearrangements) are detected at baseline, on day 15 and before surgery.

SUMMARY:
This study is to explore the markers in early prediction of the efficacy of pre-operative pertuzumab plus trastuzumab (PH) combined with chemotherapy for early stage or locally advanced human epidermal growth factor receptor-2 (HER-2) positive primary breast cancer.

DETAILED DESCRIPTION:
This study is to evaluate the correlation between early changes in multiple markers and pathological complete response in breast and lyphm nodes (tpCR) in patients with HER2-positive breast cancer receiving carboplatin, docetaxel and trastuzumab plus pertuzumab (TCHP) pre-operatively. The markers would be examined by gene expression assays, fluorodeoxyglucose positron emission tomography (18F-FDG-PET), 68 Ga-Affibody HER-2 Imaging PET, and organoid drug sensitivity test. Approximately 94 patients were treated with PH-based neoadjuvant therapy followed by surgery, and would complete 1 year of PH-based regimen in the adjuvant setting. The primary endpoint is the percent change of SUVmax from baseline to Day 15 (after the first cycle of anti HER-2 targeting drug treatment) on FDG PET and HER-2 imagining PET in correlation with pathological complete response (pCR) in patients treated with preoperative pertuzumab and trastuzumab. pCR was defined as no viable invasive cancer in breast and axilla by local pathology review.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, presenting for the first time with operable breast cancer, who had not received any previous treatment for an invasive malignancy.
2. Primary tumor greater than (>) 2 cm in diameter.
3. Age ≥ 18 years and < 70 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (</=) 1.
5. Baseline left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 55%
6. Availability of tumor tissue specimen after surgery.
7. Participants agree to undergo a core needle biopsy for genomic testing and organoid drug sensitivity assay.
8. Histologically proven diagnosis of breast cancer.
9. Patients have HER2-positive disease. HER2-positive disease was defined as follows: disease which overexpresses HER-2 by immunohistochemistry (IHC) 3+ and/or has HER2 amplification according to fluorescence in situ hybridization (FISH).
10. Had hormonal receptors (ER and PgR) assessed.
11. Signed informed consent.
12. Able to comply with the protocol.

Exclusion Criteria:

1. Metastatic disease (Stage IV) or bilateral breast cancer.
2. Any previous systemic therapy (including chemotherapy, immunotherapy, HER2 targeted agents, and antitumor vaccines) for cancer, or radiation therapy for cancer.
3. Prior breast or non-breast malignancy within 5 years prior to study entry.
4. Inadequate bone marrow, renal, or liver function
5. History or evidence of cardiovascular condition
6. Severe, uncontrolled systemic disease
7. Participants with poorly controlled diabetes or with evidence of clinically significant diabetic vascular complications.
8. Pregnancy or breast-feeding women.
9. Participants who received any investigational treatment within 4 weeks of study start.
10. Participants with known infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
11. Current chronic daily treatment with corticosteroids (dose >10 mg methylprednisolone or equivalent [excluding inhaled steroids]).
12. Known hypersensitivity to any of the study drugs or excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Standardized Uptake Value (SUV) on Positron Emission Tomography and Change in Gene Expression With Response | From baseline to day 15
  Change in SUVmax from baseline to Day 15 on 18-FDG PET and 68Ga-Affibody HER-2 Imaging PET in correlation with pathological complete response (pCR) in patients treated with preoperative pertuzumab/trastuzumab.

SECONDARY OUTCOMES:
Pathologic complete response in the breast and lymph nodes (ypT0/Tis ypN0) | Immediately after the surgery
  To determine whether the composite markers can predict pathologic complete response in the breast and lymph nodes in HER-2 positive breast cancer with PH combination with chemotherapy adjuvant therapy. Defined as the absence of any invasive component in the resected breast specimen and all resected lymph nodes following completion of neoadjuvant therapy (ypT0/Tis ypN0).
Invasive disease-free survival (iDFS) (excluding Second Primary Non-Breast Cancer [SPNBC]) | Following surgery until Year 5
  To determine the correlation between the composite markers and invasive disease free survival in HER-2 positive breast cancer patients receiving docetaxel, carboplatin, and trastuzumab plus pertuzumab pre-operatively. iDFS event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence; ipsilateral local-regional invasive breast cancer recurrence; distant recurrence; death attributable to any cause; contralateral invasive breast cancer. All SPNBCs and in situ carcinomas (including ductal carcinoma in situ [DCIS] and lobular carcinoma in situ [LCIS]) and non-melanoma skin cancer were excluded as an event.
iDFS (including SPNBC) | Following surgery until Year 5
  The iDFS event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence; ipsilateral local-regional invasive breast cancer recurrence; distant recurrence; death attributable to any cause; contralateral invasive breast cancer; SPNBC (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Overall survival (OS) | Following surgery until Year 5
  To determine the correlation between the composite markers and overall survival in HER-2 positive breast cancer patients receiving docetaxel, carboplatin, and trastuzumab plus pertuzumab pre-operatively. Percentage of participants who died due to any cause is reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code